CLINICAL TRIAL: NCT07182058
Title: Virtual Remote Assessment of Transcranial Electrical Stimulation for Parkinson's Disease Motor Symptoms
Brief Title: Virtual tES Device Treatment for Parkinson's Disease Motor Symptoms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U: The Mind Company (Industry)
Responsible Party: Principal Investigator, Mohammed Abouelsoud, CEO, Neurotechnologist, U: The Mind Company
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-PD-USA-2025-001
Record Dates: First submitted 2025-09-16; First posted 2025-09-19 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Tremor; Rigidity; Dyskinesia; Bradykinesia; Gait Dysfunction
MeSH Terms: conditions — Parkinson Disease; Tremor; Muscle Rigidity; Dyskinesias; Hypokinesia

STUDY DESIGN:
Intervention Model Description: Single-arm study where all participants receive active transcranial electrical stimulation treatment with the Sphere V3.0 device. No control or placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active Treatment Arm (Experimental): All participants receive active transcranial electrical stimulation treatment using the Sphere V3.0 device. Treatment consists of 13-minute daily sessions Monday through Friday for 3 weeks (15 total sessions), followed by 3 weeks of follow-up monitoring without device use. The device delivers amplitude-modulated transcranial pulsed random noise stimulation (am-tPRNS) with current intensity up to 4mA through a 4-electrode array placed on the scalp targeting motor cortex regions.
  Interventions: Device: Transcranial Electrical Stimulation Device

INTERVENTIONS:
Device: Transcranial Electrical Stimulation Device — The Sphere V3.0 is a non-invasive transcranial electrical stimulation device that delivers amplitude-modulated transcranial pulsed random noise stimulation (am-tPRNS).

SUMMARY:
This study tests a new, non-invasive brain stimulation device called Sphere V3.0 to help improve movement problems in people with Parkinson's disease. The device delivers gentle electrical signals to the scalp using small electrodes placed on the head.

Participants will use the device at home for 13 minutes each weekday (Monday through Friday) for 3 weeks, then be monitored for another 3 weeks without treatment. The entire study lasts 6 weeks and is conducted virtually through video calls and online assessments.

The investigators will measure changes in Parkinson's symptoms using standard rating scales and video recordings of movement tasks like walking and hand tremor tests. Participants will also record videos of their movements at home using their smartphone or computer.

The study includes 30 adults aged 18-80 who have been diagnosed with Parkinson's disease and have stable medication for at least 4 weeks. Participants must have reliable internet access and be able to follow the treatment schedule.

The main goal is to see if this brain stimulation treatment can reduce motor symptoms like tremor, stiffness, and slowness of movement. The investigators will also check if any improvements last after treatment ends and monitor for any side effects.

All participants receive the active device treatment - there is no placebo group. The device has been tested in over 250 people in previous studies with no serious adverse events reported

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Transcranial electrical stimulation (tES) represents a promising non-invasive approach for treating Parkinson's disease motor symptoms. The Sphere V3.0 device utilizes amplitude-modulated transcranial pulsed random noise stimulation (am-tPRNS) with randomized timing parameters to target motor cortex regions. Previous clinical experience with this technology includes over 250 participants across multiple studies with over 30,000 hours of treatment data and no adverse events recorded.

VIRTUAL STUDY DESIGN:

This fully remote study leverages HIPAA-compliant telehealth platforms to conduct all assessments and monitoring virtually. Participants receive the device via mail with comprehensive training materials and video tutorials. Virtual onboarding includes supervised device setup and electrode placement training via video call.

DEVICE SPECIFICATIONS:

The Sphere V3.0 employs a 4-electrode array configuration with 3D-printed dry electrodes and dual-channel programmability. Stimulation parameters include pulse duration of 450-650ms (randomly varied), inter-pulse intervals of 45-65ms, phase durations of 4.5-5.5 seconds, and current intensity up to 4mA maximum. Safety features include current limiting circuitry, automatic shutoff if skin contact is compromised, and biocompatible electrode materials.

COMPUTER VISION ANALYSIS:

Dual video protocols collect standardized movement assessments for objective analysis. Protocol A focuses on computer vision analysis with specific camera positioning for tremor (top-down view with white tablecloth) and gait assessment (perpendicular and end-on camera angles). Protocol B provides standard clinical videos for potential future MDS-UPDRS scoring. All videos are collected at consistent times, preferably before 9 AM.

SAFETY MONITORING:

Comprehensive remote safety monitoring includes weekly digital diary submissions, 24/7 emergency hotline support, and predefined escalation pathways. Level 1 events (mild headache, slight skin irritation) are documented in daily diaries. Level 2 events (persistent symptoms) require immediate hotline contact. Level 3 events (severe symptoms) mandate device cessation and emergency medical evaluation.

DATA COLLECTION SYSTEMS:

All data is collected through encrypted, HIPAA-compliant electronic data capture systems with secure cloud-based storage. Device usage metrics are transmitted in real-time to study coordinators. Video uploads utilize automated processing for standardized analysis.

REGULATORY CLASSIFICATION:

This study operates under Non-Significant Risk (NSR) device classification, providing expedited regulatory pathway while maintaining full IRB oversight and FDA compliance standards.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-80 years with confirmed diagnosis of Parkinson's Disease
* Hoehn & Yahr stages 1-4
* Stable medication regimen for 4+ weeks prior to enrollment
* Reliable internet access and telehealth capability
* Ability to provide informed consent
* Willingness to comply with treatment protocols and follow-up procedures

Exclusion Criteria:

* Metallic head/neck implants (excluding dental fillings)
* Pregnancy or nursing status
* Severe skin conditions at electrode placement sites
* History of epilepsy or seizures (unless technology specifically indicated)
* Recent stroke or traumatic brain injury (within 6 months)
* Severe cognitive impairment preventing treatment understanding
* Any neurological disorders contraindicating transcranial electrical stimulation
* Current participation in other clinical trials
* Inability to commit to full treatment and follow-up schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in MDS-UPDRS Part III Motor Scores | Baseline to Week 3 (end of treatment)
  Change from baseline to end of treatment in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III motor examination scores. The MDS-UPDRS Part III assesses motor signs of Parkinson's disease including tremor, rigidity, bradykinesia, and postural instability. Scores range from 0-132 with higher scores indicating worse motor function. All assessments conducted by qualified medical personnel including physicians, certified research coordinators, or trained clinical research assistants under physician supervision.

CONTACTS AND LOCATIONS:
Locations (1):
- U LLC Headquarters, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided